CLINICAL TRIAL: NCT02479347
Title: A Randomized, Blinded, Single Center Study to Assess the Incidence of Surgical Site Infections in Breast Cancer Surgery After Preoperative Skin Preparation With Chlorhexidine 2% in Alcohol 70% (CHLORAPREP ®) Versus 10% Povidone-iodine
Brief Title: Wound Infections in Breast Cancer Surgery After Preoperative Skin Preparation With Chlorhexidine vs. Povidone-iodine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: INT-81/12; 2012-002460-27 (EudraCT Number)
Record Dates: First submitted 2015-06-15; First posted 2015-06-24 (Estimated); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Wound Infection; Breast Neoplasms
Keywords: General surgery; Postoperative
MeSH Terms: conditions — Wound Infection; Breast Neoplasms | interventions — Chlorhexidine; Povidone-Iodine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chloraprep (Experimental): Preoperative skin preparation with chlorhexidine 2% in alcohol 70% solution
  Interventions: Drug: Chlorhexidine
- Povidone-iodine (Active Comparator): Preoperative skin preparation with povidone-iodine 10% solution
  Interventions: Drug: Povidone-Iodine

INTERVENTIONS:
Drug: Chlorhexidine — Preoperative skin preparation with tinted chlorhexidine gluconate 2% in 70% isopropyl alcohol administered with single-dose applicator
  Other Names: Chloraprep (Carefusion)
  Arms: Chloraprep
Drug: Povidone-Iodine — Preoperative skin preparation with povidone-iodine 10% aqueous solution
  Other Names: Betadine
  Arms: Povidone-iodine

SUMMARY:
The development of surgical site infections (SSI) in clean-contaminated surgery is regarded as being preventable. Known to be effective in the prevention of surgical site infection are the adequate sterilization of the surgical instruments, asepsis during operation, antibiotic prophylaxis where indicated, and certainly the preparation of the skin at the incision site, since the patient's skin is the principal source of bacterial contamination of the wound. This study aims to investigate the efficacy in prevention of surgical site infection in clean surgery, using two different standardized methods of skin preparation: povidone-iodine 10% aqueous solution from 1.5 liter bulk bottle, versus tinted 2% chlorhexidine in 70% isopropyl alcohol in a single-dose applicator. To reduce the variables involved, a single-center study will enroll a homogeneous population, undergoing breast cancer surgery.

DETAILED DESCRIPTION:
The development of surgical site infections (SSI) in clean-contaminated surgery is regarded as being preventable. Known to be effective in the prevention of surgical site infection are the adequate sterilization of the surgical instruments, asepsis during operation, antibiotic prophylaxis where indicated, and certainly the preparation of the skin at the incision site, since the patient's skin is the principal source of bacterial contamination of the wound. Products generally used for preoperative preparation of the skin are iodophores (povidone-iodine), and products containing alcohol and/or chlorhexidine.

To date, in the literature there are quite a number of case studies, but only few randomized controlled trials (RCTs) that compare different methods of preparation of the skin at the site of surgery. Only recently a major study comparing between 2 modes of skin preparation before surgery has been performed and published, and at least 2 systematic reviews of various methods can be found. At present, the use of chlorhexidine in alcohol is seen to be more effective than povidone-iodine in the prevention of surgical site infection, but the data derived from the available studies are not sufficient to definitely support a change in the daily practice, and quantitative evaluation of pharmaco-economics implications are still missing.

This study aims to investigate the efficacy in prevention of surgical site infection in clean surgery, using two different standardized methods of skin preparation: povidone-iodine 10% aqueous solution from 1.5 liter bulk bottle, versus tinted 2% chlorhexidine in 70% isopropyl alcohol in a single-dose applicator. To reduce the variables involved, a single-center study will enroll a homogeneous population, undergoing breast cancer surgery.

The patients included in this study will be randomized according to the week in which they will receive surgical treatment. The investigators expect this approach to be easier to manage within this study. The randomly assigned treatment will be weekly communicated to the chief nurse of the operating theatre who will supply the proper disinfectant without any other role in the study.

All patients will be scheduled for at least one follow up visit after about 2 weeks after surgery. All patients have access to more follow up visits, if needed, and will be asked to report all kind of wound complications.

The wound assessment will be made by persons not aware of the treatment arm the patient was assigned to, and a defined protocol assessment, based on Centers for Disease Control and prevention (CDC) definitions, which provides the following classification:

1. absence of infection;
2. superficial wound infection;
3. deep wound infection. The final follow-up visit during which the patient will be evaluated will be conducted at 30 days (for patients without insertion of prosthesis / expander) and at 180 days (for patients with the insertion of implants / expander).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing breast surgery at the Fondazione IRCCS National Cancer Institute in Milan (Italy), with or without reconstructive surgery / prosthesis or expander insertion
* Acceptance of the procedures of the protocol
* Signature of informed consent for the study

Exclusion Criteria:

* Refusal of the patient
* Age < 18 years
* Pregnancy
* Patients undergoing abdominal DIEP flap reconstruction
* Allergy to one of the disinfectants;
* Pre-existing infection in any body site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2158 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Incidence of wound infection after surgery (composite outcome) | 30 days after surgery without breast implant and 180 days after surgery with implant
  Overall incidence of surgical site infections after surgery

SECONDARY OUTCOMES:
Incidence of deep surgical site infection after surgery without implant | 30 days after surgery
  Overall incidence of surgical site infections after surgery without implant
Incidence of deep surgical site infection after surgery with implant | 180 days after surgery
  Overall incidence of surgical site infections after surgery with implant
Risk factors for surgical site infection evaluation | 30 and 180 days after surgery
  Multivariate analysis of risk factors: presence or absence of implant, previous chemotherapy treatment, previous radiotherapy treatment, American Society Association class > 2, length of surgery > 2 hours, body mass index > 35, diabetes mellitus
Analysis of extra-cost indicators | 180 days after surgery
  Record of number of additional hospital admission due to wound infection; Length of hospital stay; Need for additional surgery due to wound infection;Days of additional antibiotic therapy due to wound infection

OTHER OUTCOMES:
Cost-effective analysis | 180 days after surgery
  Cost-effective analysis if one treatment proves significantly superior to the other

CONTACTS AND LOCATIONS:
Overall Officials: Martin Langer, Prof, Study Chair — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Mi, Italy

REFERENCES:
- [Background] Mangram AJ, Horan TC, Pearson ML, Silver LC, Jarvis WR. Guideline for prevention of surgical site infection, 1999. Hospital Infection Control Practices Advisory Committee. Infect Control Hosp Epidemiol. 1999 Apr;20(4):250-78; quiz 279-80. doi: 10.1086/501620. No abstract available. PMID 10219875
- [Background] Darouiche RO, Wall MJ Jr, Itani KM, Otterson MF, Webb AL, Carrick MM, Miller HJ, Awad SS, Crosby CT, Mosier MC, Alsharif A, Berger DH. Chlorhexidine-Alcohol versus Povidone-Iodine for Surgical-Site Antisepsis. N Engl J Med. 2010 Jan 7;362(1):18-26. doi: 10.1056/NEJMoa0810988. PMID 20054046
- [Background] Lee I, Agarwal RK, Lee BY, Fishman NO, Umscheid CA. Systematic review and cost analysis comparing use of chlorhexidine with use of iodine for preoperative skin antisepsis to prevent surgical site infection. Infect Control Hosp Epidemiol. 2010 Dec;31(12):1219-29. doi: 10.1086/657134. Epub 2010 Oct 22. PMID 20969449
- [Background] Noorani A, Rabey N, Walsh SR, Davies RJ. Systematic review and meta-analysis of preoperative antisepsis with chlorhexidine versus povidone-iodine in clean-contaminated surgery. Br J Surg. 2010 Nov;97(11):1614-20. doi: 10.1002/bjs.7214. PMID 20878942